CLINICAL TRIAL: NCT07223372
Title: Treatment Patterns and Characteristics of Patients Receiving Androgen Receptor Pathway Inhibitors in a Real-world Setting in -Australia: A Retrospective Prescriptions Data Study (TARA)
Brief Title: An Observational Study to Learn More About How Medicines That Block Male Hormones Are Used in People With Prostate Cancer in Australia
Acronym: TARA
Status: Not yet recruiting | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 23084
Record Dates: First submitted 2025-10-24; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Hormonesensitive Prostate Cancer (mHSPC)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: Patients who received darolutamide
- Cohort 2: Patients who received enzalutamide
- Cohort 3: Patients who received apalutamide
- Cohort 4: Patients who received abiraterone/methylprednisolone

SUMMARY:
This is a retrospective, observational study looking at real-world prescription data in Australia. The study focuses on adult men with metastatic hormone-sensitive prostate cancer (mHSPC), a type of prostate cancer that has spread but still responds to hormone therapy. The main goal is to understand the treatment patterns, characteristics, and outcomes for patients who are receiving a class of drugs called Androgen Receptor Pathway Inhibitors (ARPIs), such as darolutamide, enzalutamide, apalutamide, or abiraterone. These drugs are often used in combination with standard Androgen Deprivation Therapy (ADT). The research will use two large, de-identified Australian prescription databases: the Pharmaceutical Benefits Scheme (PBS) and the NostraData retail pharmacy dataset. By analyzing this information, the study aims to describe how these treatments are being used over time, including what proportion of patients receive doublet therapy (ARPI + ADT) or triplet therapy (ARPI + ADT + docetaxel chemotherapy). It will also describe the characteristics of the patients receiving these therapies, such as their age and location. Secondary goals include understanding how well patients adhere to their prescribed ARPI treatment and tracking any changes in medication dosage over time. Since the study uses existing, anonymized data, there is no direct contact with patients and individual patient consent is not required. The findings will provide valuable real-world insights into the use of ARPIs in Australia, which can help inform clinical practice and improve care for men with mHSPC.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with evidence of mHSPC at any point during the study period.
* At least one dispensing of darolutamide or enzalutamide or apalutamide or abiraterone acetate/methylprednisolone, initiated for the first time during the patient identification period for mHSPC
* Age ≥18 years at index date.
* At least 12 months of data prior to index date (a sensitivity analysis will also be conducted using 6 months pre-index period)
* At least 3 months of data after index date (a sensitivity analysis will also be conducted using 6 months post-index period)

Exclusion Criteria:

* Evidence of prior use of ARPI, including darolutamide, enzalutamide, apalutamide, or abiraterone/methylprednisolone, before the index date
* Evidence of castration resistant prostate cancer (CRPC), either metastatic or nonmetastatic, before or on the index date, proxied by timing of medications in use.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: This study is a retrospective, observational analysis of prescription data collected in Australia from real-world data sources: the Pharmaceutical Benefits Scheme (PBS) 10% sample data and NostraData. Target population were adult male mHSPC patients who initiated ARPI therapy within the study period, either in doublet or triplet therapy with ADT and/or docetaxel.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-11-07 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number and proportion of patients taking each ARPI as a percentage of total study population. | Retrospective analysis from December 2022 to June 2025
Demographic characteristics of mHSPC patients | Retrospective analysis from December 2022 to June 2025

SECONDARY OUTCOMES:
Proportion of days covered (PDC) to understand adherence | Retrospective analysis from December 2022 to June 2025
  Evaluation of treatment adherence from treatment initiation using a proportion of days covered (PDC) analysis. PDC is calculated as the number of days with medication available divided by the total number of days in the observations period, starting from ARPI (Andorgen receptor pathway inhibitor) initiation
Starting dose and change in dose over time | Retrospective analysis from December 2022 to June 2025

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.